CLINICAL TRIAL: NCT01707173
Title: Improving the Self-Efficacy of African American Parents in Infant Supine Sleep
Acronym: PrAAIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Kathryn Moseley, MD, MPH, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1R01HD064770-01A1 (NIH); HUM00048679 (Other: University of Michigan); R01HD064770 (NIH)
Record Dates: First submitted 2012-10-11; First posted 2012-10-16 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: African American Infant Sleep Beliefs and Practices
Keywords: SIDS
MeSH Terms: conditions — Sudden Infant Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Education (Other): Control group participants will receive standard educational materials published by the CDC or American Academy of Pediatrics as an intervention along with a generic infant safety DVD
  Interventions: Behavioral: Standard Education
- Tailored education (Experimental): Parents/caregivers will receive educational materials tailored to their specific beliefs and barriers about infant supine sleep along with a DVD detailing standard guidelines along with specific solutions and facilitators to infant supine sleep as the intervention.
  Interventions: Behavioral: Tailored education

INTERVENTIONS:
Behavioral: Tailored education — Using information gleaned from interviews, educational print materials tailored to the participant's beliefs about infant safe sleep practices, will be mailed to the participants home at 2 separate times over a 6 month period along with a culturally relevant DVD with safe sleep information
  Arms: Tailored education
Behavioral: Standard Education — Participants will receive currently available publications about infant sleep from the American Academy of Pediatrics and the AAP at 2 separate times over a 6 month period along with a generic DVD about infant safety practices
  Arms: Standard Education

SUMMARY:
This is a research study of African American parents/caregivers of newborns. The purpose of this research study is to learn what type of educational materials about infant safety and safe infant sleep are most effective and acceptable to parents and caregivers. The investigators will compare the responses of parents who receive enhanced materials to the responses of parents who receive the ordinary materials that are currently in use.

DETAILED DESCRIPTION:
The goal of the proposed research is to determine whether a tailored multi-media mailed intervention is superior to standard non-tailored print brochures along with a generic DVD in increasing the prevalence of African American infant supine sleep during the first six months of life.

ELIGIBILITY:
Inclusion Criteria:-

- Self-identified AA adult parents and primary caregivers (≥ 18 years of age) of newborns ≤ four weeks old at the time of the infant's first office visit to the pediatrician.

Exclusion Criteria:

* Foster parents and temporary guardians:
* Prior study participants:
* Parents without a reliable phone number:
* Parents without ready access to a DVD player: an ownership of a DVD player,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 735 (Actual)
Dates: Start 2012-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Infant's usual sleep position per parental report | Change in position from study entry to infant ages 3 months and to six months; change in position from infant ages 3 months to 6 months
Infants position for last night's sleep per parental report | Change in position from study entry to infant ages 3 months and six months; change in position from infant age 3 months to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn L Moseley, MD, MPH, Principal Investigator — University of Michigan
Locations (1):
- Child Health Evaluation and Research Unit, University of Michigan, Ann Arbor, Michigan, United States